CLINICAL TRIAL: NCT00477386
Title: Phase I/II Trial of Decitabine as a Sensitizer to Carboplatin in Platinum Resistant Recurrent Ovarian Cancer
Brief Title: Trial of Decitabine as a Sensitizer to Carboplatin in Platinum Resistant Recurrent Ovarian Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Indiana University (Other)
Collaborators: Eisai Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0704-07 IUCRO-0185
Record Dates: First submitted 2007-05-21; First posted 2007-05-23 (Estimated); Results first posted 2014-09-25 (Estimated); Last update posted 2014-09-25 (Estimated); Status verified 2014-09

CONDITIONS: Ovarian Cancer
Keywords: recurrent ovarian cancer; platinum resistant; decitabine
MeSH Terms: conditions — Ovarian Neoplasms | interventions — Decitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Carboplatin combined with Decitabine (Experimental): Decitabine at escalating dose levels will be given X 5 days followed by Carboplatin given on Day 8.
  Interventions: Drug: decitabine

INTERVENTIONS:
Drug: decitabine — Decitabine dose will be escalated as follows.
  Dose level 1: 10mg/m2 IV QD X 5 days Dose level 2: 20mg/m2 IV QD X 5 days Dose level -1: Carboplatin AUC 4.
  Other Names: 5-aza-dCyd; deoxyazacytidine; dezocitidine; Dacogen

SUMMARY:
Based on these pre-clinical data, which were generated by our group, the investigators propose to test in a phase I/II clinical trial the following hypothesis: demethylation induced by decitabine results in re-sensitization to platinum in recurrent ovarian cancer.

To test this hypothesis, the investigators will treat patients with recurrent ovarian cancer platinum resistant (recurrence within 6 months from platinum therapy) or platinum-refractory (no response to platinum) with a combination consisting of decitabine and carboplatin.

This will be an institutional open label phase I/II trial to determine the safety and the biologic activity of the Decitabine/Carboplatin combination.

The investigators will determine whether Carboplatin can be safely combined with Decitabine, the optimal dose schedule and the investigators will define whether at this dosage, the regimen is biologically active (i.e. induces demethylation of target genes).

In the second part of the trial, the investigators will determine the clinical activity of the combination in a population of patients with platinum-resistant ovarian cancer.

DETAILED DESCRIPTION:
Decitabine at escalating dose levels will be given IV X 5 days followed by Carboplatin given IV on Day 8 at a dose corresponding to an area under curve (AUC) of 5. The maximum dose of Decitabine (20 mg/m2) is based on the results of the myelodysplastic syndrome (MDS) clinical trial that demonstrated biological and clinical efficacy at this dose (15-17). It is recognized that higher doses of decitabine can be administered, myelotoxicity being the most significant adverse event. This protocol will assess the lower less toxic but biologically active dose.

Decitabine dose will be escalated as follows.

Dose level -1: 5 mg/m2 IV per day (QD) X 5 days Dose level 1: 10mg/m2 IV QD X 5 days Dose level 2: 20mg/m2 IV QD X 5 days

Each cycle will consist of 28 days, with delays to allow blood count recovery. Correlative blood draws will occur on Day1 (baseline) and on Day 8 before Carboplatin for cycle 1 and 2.

The escalation phase will follow the standard 3+3 design. That is, patients will be accrued to each dose level in cohorts of up to 3-6 patients. Escalation will continue until a DLT is observed, the highest dose-level is reached, or medical judgment indicates. The goal of the phase I cohort is to ensure the safety and tolerability of the combination, not to define the maximum tolerated dose.

An initial 3 patients will be enrolled at dose level 1. If all 3 patients in dose level 1 complete 4 weeks of therapy without dose limiting toxicity (DLT), the study will proceed to enroll 3 patients at dose level 2. If all 3 patients in dose level 2 complete 4 weeks of therapy without DLT, we will accrue 3 more to ensure that only 0 or 1 of 6 have a DLT and then proceed to the phase II cohort. As dose level 2 represents full doses of both agents, there will be no further dose escalation beyond dose level 2.

ELIGIBILITY:
Inclusion Criteria:

- Have recurrent epithelial ovarian cancer, primary peritoneal carcinomatosis or fallopian tube cancer. - Have platinum-resistant (recurrence within 6 months of a platinum-containing regimen) or platinum refractory (progression while on platinum) disease - Have measurable disease according to RECIST or detectable disease. o Measurable disease is defined as the presence of at least one uni-dimensionally measurable lesion greater than or equal to 20 mm by conventional techniques, including palpation, plain x-ray, CT scan or MRI, or greater than or equal to 10 mm by spiral CT scan. o Detectable disease is defined in a patient as one who does not have measurable disease but has at least one of the following conditions: 1) Baseline values of cancer antigen 125 (CA-125) at least twice the upper limit of normal; 2) Ascites and/or pleural effusion attributed to tumor; 3) solid and/or cystic abnormalities on radiographic imaging that do not meet RECIST definitions for target lesions. - >/= 18 years of age. - Give written, informed consent for participation in the protocol. - Be at least 4 weeks from last treatment to allow recovery from prior toxicity (with the exception of hormonal therapy, where a 1-week wash-out period and radiation therapy where a 3-week wash-out period are sufficient). Patients coming off experimental therapy with biological agents not expected to cause myelotoxicity should have been off treatment for at least 3 weeks as wash-out period. - Have had disease that has progressed within 6 months platinum-based chemotherapeutic regimen. - Have no history of platinum allergy. - Have a negative serum pregnancy test prior to the study entry and be practicing an effective form of contraception if hysterectomy and/or oophorectomy were not part of the prior treatment. It is expected that the overwhelming majority of ovarian cancer patients would have had hysterectomy and oophorectomy as part of the original surgery. - Have Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1. - Have acceptable organ function, as evidenced by laboratory data: o Aspartate aminotransferase and alanine aminotransferase less than 2.5 times upper limit of normal (ULN) o Direct bilirubin less than 1.5 times ULN o Alkaline phosphatase less than 2.5 times ULN o Absolute neutrophil count greater than or equal to 1500 cells/mm3 o White cell blood count greater than 3000cells/mm3 o Hemoglobin greater than or equal to 9.0 g/dL (can be post-transfusion) o Platelets greater than 100,000/mm3 (can not be post-transfusion) o Creatinine levels less than 1.5 times ULN

Exclusion Criteria:

- Not have participated in any clinical trial involving conventional or investigational drugs or devices within the previous 3 weeks. - Not have grade 2 or greater neuropathy. - Have no additional active cancer in addition to the epithelial ovarian cancer within the last 5 years, with the exception of superficial skin cancer (basal cell or squamous cell skin carcinoma), carcinoma in situ of the cervix, Stage I endometrial cancer with less than 50% invasion of the myometrium, or other adequately treated Stage I or II cancer in complete remission. - Be free of active infection requiring antibiotic treatment. - Not have an additional uncontrolled serious medical condition or psychiatric illness. - Not have an immune deficiency and be receiving combination anti-retroviral therapy - Not have known brain metastases, as progressive neurologic dysfunction may develop, that would confound the evaluation of neurologic and other adverse events. - Absence of uncontrolled hypertension, arrhythmia, congestive heart failure or angina. Patients who have had a myocardial infarction or cardiac surgery should be at lease 6 months from the event and free of active symptoms.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2007-07; Primary Completion 2011-05 (Actual); Study Completion 2013-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniela Matei, MD, Principal Investigator — Indiana University
Locations (1):
- Indiana University Cancer Center, Indianapolis, Indiana, United States

REFERENCES:
- [Result] Matei D, Fang F, Shen C, Schilder J, Arnold A, Zeng Y, Berry WA, Huang T, Nephew KP. Epigenetic resensitization to platinum in ovarian cancer. Cancer Res. 2012 May 1;72(9):2197-205. doi: 10.1158/0008-5472.CAN-11-3909. PMID 22549947
- [Result] Fang F, Balch C, Schilder J, Breen T, Zhang S, Shen C, Li L, Kulesavage C, Snyder AJ, Nephew KP, Matei DE. A phase 1 and pharmacodynamic study of decitabine in combination with carboplatin in patients with recurrent, platinum-resistant, epithelial ovarian cancer. Cancer. 2010 Sep 1;116(17):4043-53. doi: 10.1002/cncr.25204. PMID 20564122

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Eleven patients were enrolled in the dosing finding Phase I part of the study. The Phase II dose treatment phase had 17 patients enrolled. This was in line with what had been planned.
Groups:
- Phase I Dose Finding: Decitabine at escalating dose levels will be given IV for 1 hour x 5 days followed by Carboplatin given IV for 30 minutes on Day 8 at a dose corresponding to an AUC of 5.
- Phase II: Decitabine at 10 mg/m2 will be given by IV for 1 hour x 5 days followed by Carboplatin given IV for 30 minutes on Day 8 at a dose corresponding to an AUC of 5.
Period: Overall Study
Arm/Group | Phase I Dose Finding | Phase II
Started | 11 | 17
Completed | 0 | 0
Not Completed | 11 | 17
Not completed — Adverse Event | 4 | 8
Not completed — Disease progression, relapse | 3 | 4
Not completed — Disease progression, refractory | 1 | 3
Not completed — Other | 1 | 2
Not completed — Physician Decision | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Phase I Dose Finding | Phase II | Total
Number analyzed (Participants) | 11 | 17 | 28
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 7 | 10 | 17
  >=65 years | 4 | 7 | 11
Age, Continuous [Mean (Standard Deviation); unit: Years] | 60.8 (7.8) | 61.4 (10.9) | 61.2 (9.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 17 | 28
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 11 | 17 | 28
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 11 | 17 | 28
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Phase I: Maximum Tolerated Dose (MTD) for Use in Phase II
Description: The definition of MTD will follow the standard definition of the phase I 3+3 trial concept. Dose Limiting Toxicities (DLTs) will be scored in the first cycle. Patients will be monitored for 28 days (a cycle) to determine whether a DLT is experienced for the specific dose level.
Time Frame: 28 days
Population: All patients assigned to Phase I of the study
Measure: Number; unit: mg/m2 IV QD x 5 days
Arm/Group | Phase I Dose Finding
Number analyzed (Participants) | 11
mg/m2 IV QD x 5 days | 10 (0) [0 to 0]

2. Primary Outcome: Phase II: Percent of Patients With Objective Response
Description: The percent of patients having an objective response (Complete Response or Partial Response) will be estimated with a 95% exact binomial confidence interval for the percent of patients receiving drug.
Time Frame: screening until end of study (approx 12-18 months)
Population: All Patients in Phase II of the study
Measure: Number (95% Confidence Interval); unit: percent of participants
Groups:
- Phase II Dose Treatment: Decitabine at 10 mg/m2 will be given by IV for 1 hour x 5 days followed by Carboplatin given IV for 30 minutes on Day 8 at a dose corresponding to an AUC of 5.
Arm/Group | Phase II Dose Treatment
Number analyzed (Participants) | 17
percent of participants | 35.3 [14.2 to 61.7]

3. Secondary Outcome: Phase II: Percent of Patients With Objective Response, CA125 Response or Stable Disease > 3 Months
Description: The percent of patients having an objective response (Complete Response or Partial Response) or CA125 response (Complete Response or Partial Response) or stable disease > 3 months will be estimated with a 95% exact binomial confidence interval for the percent of patients receiving drug.
Time Frame: screening until end of study (approx 12-18 months)
Population: All Patients in Phase II of the study
Measure: Number (95% Confidence Interval); unit: percent of patients
Arm/Group | Phase II Dose Treatment
Number analyzed (Participants) | 17
percent of patients | 70.6 (0) [44.0 to 89.7]

4. Secondary Outcome: Phase II: Progression Free Survival
Description: Progression free survival times will be estimated using the Kaplan-Meier method. If a patient progresses or dies, the time till that event will be used. If a patient does not progress or die on the study, the patient will be censored at the last available visit. Confidence intervals on the median will be constructed.
Time Frame: Baseline until disease progression or last visit
Population: All Patients in Phase II of the study
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Phase II Dose Treatment
Number analyzed (Participants) | 17
Months | 10.2 (0) [1.8 to 14.8]

ADVERSE EVENTS:
Time Frame: The AEs were collected from beginning of treatment until the end of study.
Groups:
- Phase I Dosing Finding: Decitabine at escalating dose levels will be given IV for 1 hour x 5 days followed by Carboplatin given IV for 30 minutes on Day 8 at a dose corresponding to an AUC of 5.
Arm/Group | Phase I Dosing Finding | Phase II
Serious Adverse Events (participants affected / at risk) | 3/11 | 4/17
Other Adverse Events (participants affected / at risk) | 10/11 | 17/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase I Dosing Finding (N=11) | Phase II (N=17)
CONSTIPATION (Gastrointestinal disorders) | 0 (0) | 1 (1)
OBSTRUCTION, GI - SMALL BOWEL NOS (Gastrointestinal disorders) | 1 (1) | 0 (0)
EDEMA: LIMB (General disorders) | 0 (0) | 1 (1)
FEBRILE NEUTROPENIA (FEVER OF UNKNOWN ORIGIN WITHOUT CLINICALLY OR MICROBIOLOGICALLY DOCUMENTED INFE (General disorders) | 1 (1) | 1 (1)
FEVER (IN THE ABSENCE OF NEUTROPENIA, WHERE NEUTROPENIA IS DEFINED AS ANC <1.0 X 10E9/L) (General disorders) | 1 (1) | 0 (0)
PAIN - HEAD/HEADACHE (General disorders) | 1 (1) | 0 (0)
PAIN - STOMACH (General disorders) | 1 (1) | 0 (0)
INFECTION WITH UNKNOWN ANC - SKIN (CELLULITIS) (Infections and infestations) | 0 (0) | 1 (1)
NEUTROPHILS/GRANULOCYTES (ANC/AGC) (Investigations) | 1 (1) | 1 (1)
PULMONARY/UPPER RESPIRATORY - OTHER (SPECIFY, __) (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
HEMORRHAGE, GI - ABDOMEN NOS (Gastrointestinal disorders) | 0 (0) | 1 (1)
LEAK (INCLUDING ANASTOMOTIC), GI - SMALL BOWEL (Gastrointestinal disorders) | 1 (1) | 0 (0)
OBSTRUCTION, GI - DUODENUM (Gastrointestinal disorders) | 1 (1) | 0 (0)
PLEURAL EFFUSION (NON-MALIGNANT) (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
THROMBOSIS/THROMBUS/EMBOLISM (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase I Dosing Finding (N=11) | Phase II (N=17)
LEUKOCYTES (TOTAL WBC) (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
LYMPHATICS - OTHER (SPECIFY, __) (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
PERICARDIAL EFFUSION (NON-MALIGNANT) (Cardiac disorders) | 0 (0) | 1 (1)
VENTRICULAR ARRHYTHMIA - VENTRICULAR TACHYCARDIA (Cardiac disorders) | 0 (0) | 1 (1)
ENDOCRINE - OTHER (SPECIFY, __) (Endocrine disorders) | 0 (0) | 1 (1)
CONSTIPATION (Gastrointestinal disorders) | 2 (2) | 9 (9)
DIARRHEA (Gastrointestinal disorders) | 2 (2) | 5 (5)
DISTENSION/BLOATING, ABDOMINAL (Gastrointestinal disorders) | 2 (2) | 3 (3)
GASTROINTESTINAL - OTHER (SPECIFY, __) (Gastrointestinal disorders) | 1 (1) | 1 (1)
HEARTBURN/DYSPEPSIA (Gastrointestinal disorders) | 0 (0) | 2 (2)
NAUSEA (Gastrointestinal disorders) | 8 (8) | 12 (12)
OBSTRUCTION, GI - SMALL BOWEL NOS (Gastrointestinal disorders) | 1 (1) | 0 (0)
TASTE ALTERATION (DYSGEUSIA) (Gastrointestinal disorders) | 0 (0) | 3 (3)
VOMITING (Gastrointestinal disorders) | 5 (5) | 5 (5)
CONSTITUTIONAL SYMPTOMS - OTHER (SPECIFY, __) (General disorders) | 0 (0) | 2 (2)
EDEMA: LIMB (General disorders) | 2 (2) | 3 (3)
FATIGUE (ASTHENIA, LETHARGY, MALAISE) (General disorders) | 5 (5) | 6 (6)
FEBRILE NEUTROPENIA (FEVER OF UNKNOWN ORIGIN WITHOUT CLINICALLY OR MICROBIOLOGICALLY DOCUMENTED INFE (General disorders) | 0 (0) | 1 (1)
FEVER (IN THE ABSENCE OF NEUTROPENIA, WHERE NEUTROPENIA IS DEFINED AS ANC <1.0 X 10E9/L) (General disorders) | 1 (1) | 3 (3)
PAIN - ABDOMEN NOS (General disorders) | 3 (3) | 7 (7)
PAIN - BACK (General disorders) | 1 (1) | 4 (4)
PAIN - BONE (General disorders) | 1 (1) | 2 (2)
PAIN - CHEST WALL (General disorders) | 0 (0) | 2 (2)
PAIN - EXTERNAL EAR (General disorders) | 0 (0) | 1 (1)
PAIN - EXTREMITY-LIMB (General disorders) | 1 (1) | 2 (2)
PAIN - HEAD/HEADACHE (General disorders) | 2 (2) | 3 (3)
PAIN - MUSCLE (General disorders) | 0 (0) | 1 (1)
PAIN - NECK (General disorders) | 0 (0) | 2 (2)
PAIN - PAIN NOS (General disorders) | 0 (0) | 3 (3)
PAIN - PELVIS (General disorders) | 0 (0) | 2 (2)
PAIN - STOMACH (General disorders) | 0 (0) | 1 (1)
ALLERGIC REACTION/HYPERSENSITIVITY (INCLUDING DRUG FEVER) (Immune system disorders) | 6 (6) | 8 (8)
INFECTION - OTHER (SPECIFY, __) (Infections and infestations) | 1 (1) | 1 (1)
INFECTION WITH NORMAL ANC OR GRADE 1 OR 2 NEUTROPHILS - BLADDER (URINARY) (Infections and infestations) | 1 (1) | 0 (0)
INFECTION WITH NORMAL ANC OR GRADE 1 OR 2 NEUTROPHILS - SINUS (Infections and infestations) | 0 (0) | 1 (1)
INFECTION WITH UNKNOWN ANC - BLADDER (URINARY) (Infections and infestations) | 0 (0) | 1 (1)
INFECTION WITH UNKNOWN ANC - LUNG (PNEUMONIA) (Infections and infestations) | 0 (0) | 1 (1)
INFECTION WITH UNKNOWN ANC - NOSE (Infections and infestations) | 0 (0) | 1 (1)
INFECTION WITH UNKNOWN ANC - SINUS (Infections and infestations) | 0 (0) | 3 (3)
INFECTION WITH UNKNOWN ANC - SKIN (CELLULITIS) (Infections and infestations) | 0 (0) | 1 (1)
INFECTION WITH UNKNOWN ANC - UPPER AIRWAY NOS (Infections and infestations) | 1 (1) | 0 (0)
ALKALINE PHOSPHATASE (Investigations) | 0 (0) | 1 (1)
HEMOGLOBIN (Investigations) | 0 (0) | 5 (5)
NEUTROPHILS/GRANULOCYTES (ANC/AGC) (Investigations) | 6 (6) | 5 (5)
PLATELETS (Investigations) | 0 (0) | 4 (4)
WEIGHT LOSS (Investigations) | 0 (0) | 1 (1)
ANOREXIA (Metabolism and nutrition disorders) | 5 (5) | 5 (5)
MAGNESIUM, SERUM-LOW (HYPOMAGNESEMIA) (Metabolism and nutrition disorders) | 0 (0) | 4 (4)
POTASSIUM, SERUM-LOW (HYPOKALEMIA) (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
FRACTURE (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
JOINT-EFFUSION (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
JOINT-FUNCTION (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
MUSCLE WEAKNESS, GENERALIZED OR SPECIFIC AREA (NOT DUE TO NEUROPATHY) - WHOLE BODY/GENERALIZED (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
MUSCULOSKELETAL/SOFT TISSUE - OTHER (SPECIFY, __) (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
COGNITIVE DISTURBANCE (Nervous system disorders) | 0 (0) | 1 (1)
DIZZINESS (Nervous system disorders) | 1 (1) | 3 (3)
MEMORY IMPAIRMENT (Nervous system disorders) | 0 (0) | 1 (1)
NEUROPATHY: CRANIAL - CN V MOTOR-JAW MUSCLES; SENSORY-FACIAL (Nervous system disorders) | 0 (0) | 1 (1)
NEUROPATHY: MOTOR (Nervous system disorders) | 0 (0) | 1 (1)
NEUROPATHY: SENSORY (Nervous system disorders) | 2 (2) | 5 (5)
SPEECH IMPAIRMENT (E.G., DYSPHASIA OR APHASIA) (Nervous system disorders) | 0 (0) | 1 (1)
SYNCOPE (FAINTING) (Nervous system disorders) | 0 (0) | 1 (1)
INSOMNIA (Psychiatric disorders) | 1 (1) | 3 (3)
MOOD ALTERATION - ANXIETY (Psychiatric disorders) | 1 (1) | 0 (0)
MOOD ALTERATION - DEPRESSION (Psychiatric disorders) | 0 (0) | 1 (1)
PSYCHOSIS (HALLUCINATIONS/DELUSIONS) (Psychiatric disorders) | 0 (0) | 1 (1)
HEMORRHAGE, GU - URINARY NOS (Renal and urinary disorders) | 1 (1) | 0 (0)
INCONTINENCE, URINARY (Renal and urinary disorders) | 0 (0) | 1 (1)
RENAL/GENITOURINARY - OTHER (SPECIFY, __) (Renal and urinary disorders) | 0 (0) | 1 (1)
URINARY FREQUENCY/URGENCY (Renal and urinary disorders) | 0 (0) | 1 (1)
HOT FLASHES/FLUSHES (Reproductive system and breast disorders) | 0 (0) | 1 (1)
LEAK (INCLUDING ANASTOMOTIC), GU - VAGINA (Reproductive system and breast disorders) | 1 (1) | 0 (0)
VAGINAL DISCHARGE (NON-INFECTIOUS) (Reproductive system and breast disorders) | 0 (0) | 1 (1)
COUGH (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 6 (6)
DYSPNEA (SHORTNESS OF BREATH) (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3)
NASAL CAVITY/PARANASAL SINUS REACTIONS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
PULMONARY/UPPER RESPIRATORY - OTHER (SPECIFY, __) (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
VOICE CHANGES/DYSARTHRIA (E.G., HOARSENESS, LOSS OR ALTERATION IN VOICE, LARYNGITIS) (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
BRUISING (IN ABSENCE OF GRADE 3 OR 4 THROMBOCYTOPENIA) (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
DERMATOLOGY/SKIN - OTHER (SPECIFY, __) (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
FLUSHING (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
HAIR LOSS/ALOPECIA (SCALP OR BODY) (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1)
PRURITUS/ITCHING (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
RASH/DESQUAMATION (Skin and subcutaneous tissue disorders) | 2 (2) | 3 (3)
RASH: ACNE/ACNEIFORM (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
SKIN BREAKDOWN/DECUBITUS ULCER (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
SWEATING (DIAPHORESIS) (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
HYPERTENSION (Vascular disorders) | 0 (0) | 1 (1)
HYPOTENSION (Vascular disorders) | 0 (0) | 1 (1)
PHLEBITIS (INCLUDING SUPERFICIAL THROMBOSIS) (Vascular disorders) | 0 (0) | 1 (1)
VASCULAR - OTHER (SPECIFY, __) (Vascular disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes